CLINICAL TRIAL: NCT01031277
Title: Centralized Gulf States Survey on the Undertreatment of Hypercholesterolemia
Brief Title: Centralized Pan-Middle East Survey on the Under-treatment of Hypercholesterolemia, Sub-study for the Gulf States
Acronym: CEPHEUS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Clinart International (Industry)
Responsible Party: MC MD, AstraZeneca Gulf States
Other Study IDs: NIS-GU-CRE-2009/1; SRP-CB-CRE-2006/01
Record Dates: First submitted 2009-12-11; First posted 2009-12-14 (Estimated); Last update posted 2011-05-25 (Estimated); Status verified 2011-05

CONDITIONS: Hypercholesterolemia
Keywords: Hypercholesterolemia; Update NCEP ATP111; Survey
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to establish the proportion of patients on lipid-lowering pharmacological treatment reaching the LDL-C goals according to the NCEP ATP III/updated 2004 NCEP ATP III guidelines, overall and by country, to establish the proportion of patients on lipid-lowering pharmacological treatment reaching the LDL-C goals according to the NCEP ATP III/updated 2004 NCEP ATP III in the following sub-populations:

* Primary/secondary prevention patients.
* Patients with metabolic syndrome (according to NCEP III definition). And to establish the proportion of patients on lipid-lowering pharmacological treatment reaching the LDL-C goals according to the Third Joint European Task Force guidelines/national guidelines, in the survey population and in the following sub-populations:

  * Primary/secondary prevention patients.
  * Patients with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Race
* On lipid-lowering drug treatment for at least 3 months, with no dose change for a minimum of 6 weeks.
* Subject must sign informed consent

Exclusion Criteria:

* Subjects who are unwilling or unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inhabitants of Gulf States visiting their cardiologist for regular follow-up of their hypercholesterolaemia treatment
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
To establish the proportion of patients on lipid-lowering pharmacological treatment reaching the LDL-C goals according to the NCEP ATP III/updated 2004 NCEP ATP III guidelines, overall and by country. | 6 months- One visit only, no follow up visits.

SECONDARY OUTCOMES:
Proportion patients on lipid-lowering drugs (LLD) reaching the LDL-C goals according to the NCEP ATP III/ updated 2004 NCEP ATP III in subgroups: Primary/secondary prevention patients; Patients with metabolic syndrome ( NCEP III). | 6 months- One visit only, no follow up visits.
Proportion patients on LLD reaching the LDL-C goals according to the Third Joint European Task Force guidelines/national guidelines, in the survey population and in sub-populations: Primary/secondary prevention patients; Patients with metabolic syndrome. | 6 months- One visit only, no follow up visits.
To identify determinants (e.g. patient and physician characteristics, country-specific guidelines or recommendations) for undertreatment of hypercholesterolemia. | 6 months- One visit only, no follow up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Wael Al Mahmeed, Study Chair — Shaikh Khalifa Medical City
Locations (1):
- Research Site, Abu Dhabi, United Arab Emirates

REFERENCES:
- [Derived] Shehab A, Al-Rasadi K, Arafah M, Al-Hinai AT, Al Mahmeed W, Bhagavathula AS, Al Tamimi O, Al Herz S, Al Anazi F, Al Nemer K, Metwally O, Alkhadra A, Fakhry M, Elghetany H, Medani AR, Yusufali AH, Al Jassim O, Al Hallaq O, Baslaib FOAS, Alawadhi M, Amin H, Al-Hashmi K, Oulhaj A. The Management of Dyslipidaemia in Patients with Type 2 Diabetes Mellitus Receiving Lipid-Lowering Drugs: A Sub-Analysis of the CEPHEUS Findings. Curr Vasc Pharmacol. 2018;16(4):368-375. doi: 10.2174/1570161115666170705153815. PMID 28677510